CLINICAL TRIAL: NCT01372891
Title: Urine Total Adiponectin and Its Isoforms Concentration in Prediction of Percutaneous Coronary Interventions Contrast Induced Nephropathy
Brief Title: Urine Adiponectin Concentration in Prediction of Contrast Induced Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: xjyy110502
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Myocardial Ischemia
Keywords: Contrast Induced Nephropathy; percutaneous coronary interventions
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum,urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients underging PCI

SUMMARY:
The present study is to determine the ability of urinary total adiponectin and its isoforms excretion in the prediction of contrast induced nephropathy (CIN) in the patients undergoing PCI.

DETAILED DESCRIPTION:
Contrast induced nephropathy (CIN) is a severe complication after percutaneous coronary intervention (PCI). CIN is responsible for approximately genic renal insufficiency and is the third cause of hospital-acquired renal failure and the injury of endothelial of renal tubule is responsible for the CIN. However markers reliably identifying CIN in the patients undergoing PCI are rare. Adiponectin is a 30-kDa adipocyte-derived vasoactive peptide closely linked to components of the metabolic syndrome. Recent study demonstrates that the quantification of urinary adiponectin excretion appears to be an independent indicator of vascular damage potentially identifying an increased risk for vascular events. Therefore, the investigators presume that the adiponectin excretion may predict the incidence of the CIN. The present study is to determine the ability of urinary total adiponectin and its isoforms excretion in the prediction of CIN in the patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 of age who are undergoing elective PCI and are able to give informed consent are eligible for study.

Exclusion Criteria:

* The end-stage renal failure
* The patients who are relieving dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls a group of patients> 18 who have ST elevation myocardial infarction (STEMI) undergoing primary PCI.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
increase in SCr 0.5 mg/dL(44.2 mol/L) from baseline | 3 days
  samples will be collected at 24, 48 and 72 hours after PCI

SECONDARY OUTCOMES:
a 25% increase in SCr from baseline | 3 days
  samples will be collected at 24, 48 and 72 hours after PCI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China